CLINICAL TRIAL: NCT05501210
Title: The Effect of Whole-Body Vibration on Patellofemoral Joint Pain After Anterior Cruciate Ligament Reconstruction
Brief Title: Vibration on Patellofemoral Joint Pain After ACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.674
Record Dates: First submitted 2022-03-22; First posted 2022-08-15 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Patellofemoral Pain
Keywords: ACLR; Patellofemoral joint; Whole Body vibration; Knee function
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into either vibration or control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WBV + PEMF Group (Experimental): Patients in "WBV + PEMF" and "WBV only" groups will be required to attend the WBV therapy session in Prince of Wales Hospital twice a week, for 8 weeks, fulfilling a total of 16 sessions. Patients in "WBV + PEMF" groups will receive PEMF after WBV session.
  Interventions: Device: WBV; Device: PEMF
- Control Group (No Intervention): Subjects in control group will perform static squat, single leg squat and lunges without vibration.
- WBV only (Active Comparator): Patients in "WBV + PEMF" and "WBV only" groups will be required to attend the WBV therapy session in Prince of Wales Hospital twice a week, for 8 weeks, fulfilling a total of 16 sessions. Patients in "WBV" groups will not receive PEMF after WBV session.
  Interventions: Device: WBV

INTERVENTIONS:
Device: WBV — Whole body vibration (WBV) therapy
  Arms: WBV + PEMF Group; WBV only
Device: PEMF — Pulsed electromagnetic fields (PEMF)
  Arms: WBV + PEMF Group

SUMMARY:
Anterior cruciate ligament (ACL) injury is a prevailing problem among sports participants, especially in non-contact sports. Studies have reported that 70-84% of ACL injuries are non-contact in nature, and movements like changing in direction while running, cutting and pivoting on a planted foot have resulted in a majority of ACL injuries. Even after ACL reconstruction (ACLR) surgeries, study has reported a 30-50% prevalence of developing patellofemoral joint (PFJ) pain in 1-2 years post-operation. Whole body vibration (WBV) therapy has been gaining attention as an effective method of training in recent years. It has been proved to have a positive effect on improving muscle strength, muscle activities, muscle power and loading during drop jump. Though duration of WBV may differ according to the effect of interest, several studies have had positive results with a 8 week WBV therapy in increasing muscle strength, proprioception, and post-ACLR knee functions. Further investigation on the underlying mechanism and possible application are to be continued to explore more possibilities with the WBV therapy.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury is a prevailing problem among sports participants, especially in non-contact sports. Studies have reported that 70-84% of ACL injuries are non-contact in nature, and movements like changing in direction while running, cutting and pivoting on a planted foot have resulted in a majority of ACL injuries. The influence of such injury can often be lifelong as it increases the patient's risk of developing degenerative musculoskeletal problems like osteoarthritis, and eventually affects the patient's quality of life. Even after ACL reconstruction (ACLR) surgeries, study has reported a 30-50% prevalence of developing patellofemoral joint (PFJ) pain in 1-2 years post-operation. The prevalence of patients developing PFJ osteoarthritis ranges from 14.8-26.5% for post-operation 2-5 years, and the percentage is even higher after more than 6 years post-operation.

Symptoms of PFJ osteoarthritis include swelling, notably reduced quadriceps strength, and pain on PFJ compression. Though the mechanism of how ACLR contributes to the development of PFJ osteoarthritis is not completely clear yet, inflammation and damage to PFJ articular cartilage and alteration of vastus medialis function, which is common after ACLR, might play a role in the development of PFJ osteoarthritis. A more than 30% decrease in quadriceps muscles strength had been reported by previous study. Decrease in size of rectus femoris, vastus medialis and vastus lateralis had also been observed. Though there was no significant difference in the vastus medialis/vastus lateralis, the decrease in strength and size of the quadricep muscles could possibly affect the stability of PFJ, increasing the chance of developing PFJ osteoarthritis.

Whole body vibration (WBV) therapy has been gaining attention as an effective method of training in recent years. More and more rehabilitation facilities have equipped the WBV machine and make this therapy more easily accessible. It has been proved to have a positive effect on improving muscle strength, muscle activities, muscle power and loading during drop jump. It has also shown effectiveness in decreasing osteoarthritic knee pain and enhancing knee function in chronic elderly knee osteoarthritis. Though the exact mechanism of the therapy is not yet very clear, it is believed that it is related to the "tonic vibration reflex". Skeletal muscles undergo small changes in muscle length during the vibration generated by the machine. It elicits the "tonic vibration reflex", activates muscle spindles and mediated neural signals. Another possible mechanism is that the vibration provides cortical stimulation and increases the corticomotor excitability. Both of them train the neuromuscular system to response faster, achieving the above-mentioned benefits.

There are different types of WBV machines, providing vertical, horizontal or pivoting vibration, and the amplitude and frequency of the vibration can be adjusted on the machine. Many studies have been conducted using different duration, amplitude and frequency of vibration. A "standard protocol" for WBV therapy is yet to be developed. Though duration of WBV may differ according to the effect of interest, several studies have had positive results with a 8 week WBV therapy in increasing muscle strength, proprioception, and post-ACLR knee functions. Further investigation on the underlying mechanism and possible application are to be continued to explore more possibilities with the WBV therapy.

Conservative and effective approaches for relieving pain are needed for knee osteoarthritis patients and, among these, pulsed electromagnetic fields (PEMF) are emerging with promising results. In vitro studies have demonstrated that PEMF therapy is effective in reducing chondrocyte apoptosis and MMP-13 expression of knee cartilage in ovariectomized rats and in favourably affecting cartilage homeostasis. PEMF was evaluated for function, a significant improvement was observed 8 weeks after initiation of treatment, and no significant association was found between the use of PEMF and the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 60
2. Unilateral ACLR
3. Persisting PFJ pain
4. Isolated symptomatic site or pathology

Exclusion Criteria:

1. Age > 60
2. Bilateral ACLR
3. Revision ACLR
4. Any rheumatological diseases
5. Previous contralateral knee injury
6. Any knee osteoarthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of The Knee injury and Osteoarthritis Outcome Score Patellofemoral subscale (KOOS-PF) | pre intervention and 8 weeks post intervention
  The KOOS-PF was developed to evaluate individuals or samples of individuals who present with anterior knee pain/patellofemoral pain and/or patellofemoral OA. It contains 11 items with 3 subscale : Stiffness, Pain, Quality of life (QOL).

SECONDARY OUTCOMES:
Isokinetic muscle strength | pre intervention and 8 weeks post intervention
  The subjects will be asked to test the muscle strength by using the isokinetic device (Biodex System 4; Biodex Medical Systems, Inc, Shirley, NY). Before testing, the subjects will be asked to have a 10-minute warm-up on a stationary bike at low intensity. By recommendation they will be asked to exert maximal concentric contraction of knee flexor and rt with the dynamometer at angular velocity of 60°/s for five times.
Muscle thickness | pre intervention and 8 weeks post intervention
  Muscle thickness of rectus femoris, vastus medialis, vastus lateralis and vastus intermedius will be assessed using ultrasound imaging. The ultrasound transducer will be placed at the muscle bellies to obtain an image of the cross-session of the muscle. The depth of the related muscle cross-session will be measured to represent the thickness of the muscle.
  Muscle thickness of rectus femoris, vastus medialis, vastus lateralis and vastus intermedius will be assessed using ultrasound imaging. The ultrasound transducer will be placed at the muscle bellies to obtain an image of the cross-session of the muscle. The depth of the related muscle cross-session will be measured to represent the thickness of the muscle.
The Numeric Pain Rating Scale (NPRS) | pre intervention and 8 weeks post intervention
  The Numeric Pain Rating Scale (NPRS):
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "the most severe pain imaginable". Scores range from 0-10 points, with higher scores indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong